CLINICAL TRIAL: NCT05202119
Title: Empower: Transcranial Direct Current Stimulation in Major Depressive Disorder: a Double-blind, Placebo-controlled, Randomized, Superiority Trial
Brief Title: Empower: tDCS for Major Depressive Disorder at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flow Neuroscience AB (Industry)
Collaborators: University of Texas (Other); University of East London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FL001
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: tDCS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and investigators are unaware of what stimulation (active or sham) the device delivers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active stimulation (Active Comparator): Active stimulation at 2mA
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation (tDCS) a non-invasive brain stimulation technique where a weak direct current (2 mA) is applied on the scalp through electrodes. The current modulates the underlying neural activity. The sessions are 30 minutes, 3-5 time a week.
  Arms: Active stimulation
Device: Sham Transcranial direct current stimulation — To blind the participants of the stimulation, a standardized sham protocol is used where the current ramped up and then down breifly in the beginning and end of each session to simulate active stimulation.
  Arms: Sham stimulation

SUMMARY:
A two-center trial to investigate whether or not active stimulation with the Flow FL-100 tDCS device is superior to sham stimulation for the treatment of major depressive disorder when used at home.

Participants perform up to 36 tDCS sessions by themselves without supervision during a blinded 10-week phase, and then 30 more sessions during an unblinded open-label phase.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years.
* Have a diagnosis of Unipolar MDD with a current depressive episode as defined by the diagnostic criteria in the Diagnostic and statistical manual of mental disorders - 5th edition (DSM-V)
* Have a Hamilton Depression Rating Score (HDRS-17) of ≥ 16.
* Have PHQ-9 of ≥10.Montgomery-Åsberg Depression Rating Scale Self-Report (MADRS-s) of ≥ 20.
* For 6 weeks prior to enrollment, are either: not taking antidepressant medication or:

are taking a stable antidepressant regimen with a stable medication source and agree to continue the same regimen throughout study participation

* If in psychotherapy, have maintained stable psychotherapy for at least 6 weeks prior to enrollment.
* Have access to a stable internet connection through which the treatment will be received.
* Have access to a smartphone or other device running Android 5.0+ or iPhone Operating System (iOS) 12+ (e.g., reasonably new iPhone/iPad or Android phone), used to using the device in their everyday life, and can capably use the study application on the device, as determined by the investigator.
* Are currently living in England/Wales (UK) or Texas (US).
* Subject is currently under the care of a psychiatrist or a primary care physician, agrees to be evaluated at regular intervals by a psychiatrist or primary care physician for the duration of study participation, and agrees to promptly inform the study staff of any change of psychiatric or mental health providers during study participation.
* Subject agrees to allow any and all forms of communication between the investigators/study staff and any healthcare provider who currently provides and/or has provided service to the patient/subject within at least two years of study enrollment.
* Subject agrees to provide the name and verifiable contact information (email and mailing addresses, mobile and land-line phone numbers, as applicable) of at least two persons ≥ age 18 (22 in the US) who reside within a 60-minute drive of the patient's residence and whom the research staff is at liberty to contact, as they deem necessary, for the duration of study participation.
* Be able to give voluntary, written informed consent to participate and have signed an Informed Consent Form specific to this study.
* Be willing and able to comply with all study procedures.
* Subject agrees to meet all of the inclusion criteria throughout their participation in the study. Otherwise, the subject will be discontinued from the study.
* Subject agrees to a Safety/Suicide Risk Management Protocol, which is intended to reduce the reduce the risk of suicide during study participation.

Exclusion Criteria:

* Are in a current state of mania, as determined by the YMRS or psychosis, as determined by the MINI.
* Are diagnosed with vitamin or hormonal deficiencies that may mimic mood disorders, as determined by the investigator.
* Are currently receiving any other interventional therapy for MDD other than a stable regimen of antidepressants or psychotherapy as defined in the inclusion criteria.
* Considered to have treatment resistant depression as defined by inadequate clinical response to 2 or more trials of antidepressants at an adequate dose and duration.
* Have a history of electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), cranial electrotherapy stimulation (CES), transcranial direct current stimulation (tDCS), deep brain stimulation (DBS), or other brain stimulation.
* Patient answers Yes to Questions 4, 5 or 6 on the Columbia Suicide Severity Rating Scale (C-SSRS) Triage and Risk Identification Screener.
* Any previous hospitilization for suicidal behavior.
* Have chronic or current severe insomnia (< 4 hours of sleep each night), or sleep apnea.
* Have any structural lesion (e.g., any structural neurological condition, or more subcortical lesions than would be expected for age or have had a stroke that affects stimulated area or connected areas) or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results, as determined by the investigator.
* Have any implant in the brain (e.g., DBS) or neurocranium, or any other active implantable medical device.
* Have any neurocranial defect.
* Have a history of epilepsy or seizures (including history of withdrawal / provoked seizures).
* Have shrapnel or any ferromagnetic material in the head.
* Have any disorder that would impair the ability to complete the study questionnaires.
* Have been diagnosed with autism spectrum disorder.
* Are actively abusing substances (<1 week prior to enrollment).
* Have a cognitive impairment (including dementia).
* Have a history of mania or psychosis.
* Are currently using any medications that affect cortical excitability (e.g., benzodiazepines, epileptics, etc.).
* Are currently experiencing symptoms of withdrawal from alcohol or benzodiazepines.
* Have been diagnosed with Parkinsonism or other movement disorder as determined by the investigator to interfere with treatment.
* Have ever taken esketamine / ketamine for treatment of depression.
* Have ever been admitted to hospital for depression.
* Have been diagnosed with obsessive-compulsive disorder (OCD), bipolar type 1 or 2 disorder, an active primary anxiety disorder, PTSD, agoraphobia, panic or personality disorder.
* Have a history of psychosurgery for depression.
* Have any history of myocardial infarction, coronary artery bypass graft (CABG), coronary heart failure (CHF), or history of other cardiac issues.
* Are currently experiencing or have a history of intractable migraines.
* Are a chronic tobacco smoker, as defined by smoking >100 cigarettes (including hand-rolled cigarettes, cigars, cigarillos, etc.) in their lifetime and has smoked every day in the last 7 days.
* If female and of child-bearing potential, currently pregnant or breastfeeding or planning to become pregnant or breastfeed any time during the study.
* Are currently a prisoner.
* Are participating concurrently in another clinical investigation or have participated in a clinical investigation within the last 90 days or intend to participate in another clinical investigation during the study.
* Have any medical condition or other circumstances, in the judgment of the investigator, that might interfere with the ability to complete follow-up visits and the self-reported MADRS-s in the app.
* Have any condition which, in the judgment of the Investigator, would preclude adequate evaluation of the device's safety and performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
HDRS-17 | 10 weeks
  Mean score change based on HDRS-17 scores of the two arms at 10 weeks compared to baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- UT Health Science Center, Houston, Texas, United States
- School of Psychology, University East London, London, United Kingdom

REFERENCES:
- [Derived] Lagerberg PJ, Woodham RD, Selvaraj S, Lajmi N, Hobday H, Sheehan G, Ghazi-Noori AR, Rizvi M, Kwon SS, Orhii P, Machado-Vieira R, Soares JC, Young AH, Fidalgo AR, Rezaei H, Fu CHY. Acceptability of active and sham home-based transcranial direct current stimulation in major depression: mixed methods qualitative analysis in a randomised controlled trial. Ann Gen Psychiatry. 2025 Dec 4;25(1):1. doi: 10.1186/s12991-025-00607-4. PMID 41345653
- [Derived] Woodham RD, Selvaraj S, Lajmi N, Hobday H, Sheehan G, Ghazi-Noori AR, Lagerberg PJ, Rizvi M, Kwon SS, Orhii P, Maislin D, Hernandez L, Machado-Vieira R, Soares JC, Young AH, Fu CHY. Home-based transcranial direct current stimulation treatment for major depressive disorder: a fully remote phase 2 randomized sham-controlled trial. Nat Med. 2025 Jan;31(1):87-95. doi: 10.1038/s41591-024-03305-y. Epub 2024 Oct 21. PMID 39433921

DOCUMENTS (1):
  • Study Protocol (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT05202119/Prot_000.pdf